CLINICAL TRIAL: NCT07264751
Title: The Effect of a Single Training Session on Changes in Inflammatory, Hormonal, and Metabolic Markers in Athletes.
Status: Completed | Type: Observational
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Anna Kasperska, Principal Investigator, Poznan University of Physical Education
Other Study IDs: AKS wrestlers
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Training; Inflammation Biomarkers; Hormone; Exercise Training
Keywords: wrestlers; catecholamines; Single training session; Inflammatory markers; Hormonal response
MeSH Terms: interventions — Physical Conditioning, Human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: physical training — The intervention consists of a standardized, high-intensity wrestling training session designed to simulate typical strength-endurance exercise performed by elite wrestlers. The session includes sport-specific drills, resistance exercises, and aerobic conditioning components appropriate for this athletic discipline. All participants will perform the session under supervision to ensure safety and adherence to the planned intensity and duration.

SUMMARY:
The study aims to assess the acute response of wrestlers to a single training session. Short-term changes in inflammatory, hormonal, and metabolic markers will be analyzed, which may reflect the development of fatigue and recovery processes following intense exercise. Participation in the study involves performing a standard training session and collecting blood samples at three time points to assess the physiological response. The results will provide a better understanding of the mechanisms of adaptation to exercise in strength and endurance athletes.

DETAILED DESCRIPTION:
The study aims to assess how wrestlers' bodies respond to a single, intense training session. The study focuses on short-term changes in markers of inflammation, the hormonal system (stress hormones, catecholamines), and the metabolic system. This enables a deeper understanding of the physiological mechanisms underlying fatigue development and post-exercise recovery.

Each participant will attend one standard training session, as outlined in the training plan. As part of the study, three venous blood samples will be collected:

* Before training - at rest, to determine baseline values;
* Immediately after training;
* 24 hours after exercise - to evaluate recovery processes.

Blood samples will be analyzed in the lab to determine:

* inflammatory markers (hsCRP, IL-6, TNF-α),
* muscle damage marker (CK),
* stress hormones (adrenaline, noradrenaline, cortisol),
* metabolic indicators (urea, creatinine, total protein, albumin, uric acid). The project does not require any additional supplementation, dietary changes, or modifications to the training plan.

Participating in the study will provide insights into your individual body's response to intense exercise, including fatigue levels, inflammation, and hormonal balance. The results can help you better tailor your training load and improve your recovery.

Participation in the study is completely voluntary. Participants may withdraw from participation at any time, without giving a reason, without any consequences. Withdrawal from the study will not affect their subsequent athletic training. All data obtained during the study will be treated confidentially and processed solely for scientific purposes. Results will be compiled in aggregate form, preventing the identification of individual participants.

The study protocol was approved by the bioethics committee.

ELIGIBILITY:
Inclusion Criteria:

* Currently engaged in regular strength-endurance wrestling training.
* Medically cleared for high-intensity exercise by a sports physician.
* Willingness to participate and provide written informed consent.
* Availability to attend the training session and all blood sampling time points (pre-training, immediately post-training, 24 hours post-training)

Exclusion Criteria:

* Presence of acute or chronic illness that may affect exercise performance or physiological response
* Recent musculoskeletal injury limiting participation in high-intensity training.
* Use of medications or supplements that may interfere with hormonal, inflammatory, or metabolic markers
* History of endocrine disorders, adrenal insufficiency, or other conditions affecting catecholamine or cortisol levels
* Inability or unwillingness to comply with study procedures.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study participants are elite wrestlers who are also members of a national-level sports club and members of the national team. All athletes have experience competing in international events. The group includes athletes who have won medals at both national and international competitions. Participants are highly trained, with extensive experience in strength-endurance wrestling disciplines, and represent the top competitive level in their sport. The study aims to evaluate acute physiological responses to a single high-intensity training session in this highly specialized discipline.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
hsCRP | 1. Before training (at rest), 2. Immediately after training, 3. 24 hours after exercise.
  highly sensitive reactive C-protein
CK | 1. Before training (at rest), 2. Immediately after training, 3. 24 hours after exercise.
  creatine kinase
TNF-alpha | 1. Before training (at rest), 2. Immediately after training, 3. 24 hours after exercise.
  tumor necrosis factor alpha
IL-6 | 1. Before training (at rest), 2. Immediately after training, 3. 24 hours after exercise.
  Interleukine-6
A | 1. Before training (at rest), 2. Immediately after training, 3. 24 hours after exercise.
  Adrenaline
Noradrenaline | 1. Before training (at rest), 2. Immediately after training, 3. 24 hours after exercise.
  Noradrenaline

SECONDARY OUTCOMES:
Kortisol | 1. Before training (at rest), 2. Immediately after training, 3. 24 hours after exercise.
  Noradrenaline
TP | 1. Before training (at rest), 2. Immediately after training, 3. 24 hours after exercise.
  total protein
Urea | 1. Before training (at rest), 2. Immediately after training, 3. 24 hours after exercise.
  Urea
Albumin | 1. Before training (at rest), 2. Immediately after training, 3. 24 hours after exercise.
  Albumin

OTHER OUTCOMES:
UA | 1. Before training (at rest), 2. Immediately after training, 3. 24 hours after exercise.
  Uric acid

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kasperska, PhD, Principal Investigator — Poznań University of Physical Education, Faculty of Sport Sciences in Gorzów Wielkopolski, Poland;
Locations (1):
- Poznań University of Physical Education, Faculty of Physical Culture in Gorzów Wielkopolski, Gorzów Wielkopolski, Polska, Poland

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to protect participant confidentiality and to meet ethical and legal standards regarding sensitive health and performance data.